CLINICAL TRIAL: NCT00214890
Title: CCTG584: Viral Dynamics and Pharmacokinetics of Tenofovir and Abacavir Monotherapy Versus the Combination Therapy of TDF-ABC in HIV-Infected Treatment Naive Patients
Brief Title: Viral Dynamics and Pharmacokinetics of Abacavir and Tenofovir
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of California, San Diego (Other)
Collaborators: Universitywide AIDS Research Program (Other); GlaxoSmithKline (Industry); University of California, Irvine (Other); University of California, Los Angeles (Other); University of Southern California (Other); Santa Clara Valley Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CCTG584
Record Dates: First submitted 2005-09-20; First posted 2005-09-22 (Estimated); Results first posted 2021-03-09 (Actual); Last update posted 2021-09-24 (Actual); Status verified 2021-09

CONDITIONS: HIV Infections
Keywords: HIV; nucleoside pharmacology; drug-drug interaction; Treatment Naive; Drug resistance; Drug pharmacokinetics
MeSH Terms: conditions — HIV Infections | interventions — Tenofovir; abacavir

STUDY DESIGN:
Intervention Model Description: This is a comparative, open-labeled study of a dual NRTI regimen, TDF + ABC, compared to ABC and TDF monotherapy administered for 7 days. Each patient will be randomized to a 7-day sequence of either ABC or TDF once-daily followed by a 35-day washout period. After completion of the monotherapy sequence all patients will then receive dual NRTI therapy of TDF + ABC for an additional 7 days. After completion of the dual NRTI sequence patients will enter the HAART treatment stage with the addition of EFV and continue on a once-daily regimen of EFV + ABC + TDF for an additional 14 days. At day 63, TDF will be stopped and 3TC will be substituted. Patients will then continue on a once-daily regimen of EFV + ABC + 3TC for an additional 46 weeks.

ARMS (2):
- Tenofovir (Active Comparator): As part of this study visit, you participants will be assigned by chance to receive either TDF alone or ABC alone
  Interventions: Drug: Tenofovir
- Abacavir (Active Comparator): As part of this study visit, you participants will be assigned by chance to receive either TDF alone or ABC alone
  Interventions: Drug: Abacavir

INTERVENTIONS:
Drug: Tenofovir — 300 mg once daily
  Other Names: (TDF)
  Arms: Tenofovir
Drug: Abacavir — 600 mg once daily
  Other Names: (ABC, Ziagen)
  Arms: Abacavir

SUMMARY:
Once-daily nucleotide/nucleoside reverse transcriptase inhibitor (NtRTI/NRTI) combinations form the backbone of many regimens. Although efficacy data exists between tenofovir and the pyrimidine analogues (i.e. lamivudine and emtricitabine), recent clinical data suggests a potential interaction between tenofovir and purine analogs (i.e. abacavir and didanosine).

Specific Aim 1: To evaluate the impact of an acyclic nucleoside phosphonate, tenofovir (TDF), on the intracellular metabolism of a purine nucleoside analog, abacavir (ABC), as a determinant of the antiviral potency of this nucleotide/nucleoside reverse transcriptase inhibitor (NtRTI/NRTI) combination.

* Hypothesis #1: ABC and TDF dosed together will have reduced antiviral activity, as measured by early plasma HIV RNA decay kinetics, than the drugs given alone.
* Hypothesis #2: ABC dosed with TDF will have reduced intracellular concentrations, as measured by the ratio of carbovir triphosphate (active metabolite of ABC) to deoxyguanosine triphosphate (endogenous nucleotide), compared to ABC given alone.

DETAILED DESCRIPTION:
The primary objectives of this study are to compare the virologic potency and pharmacology of TDF and ABC alone and in combination. Since it is not feasible or ethical to give mono or dual-therapy with these agents for prolonged intervals, this project was designed to take advantage of a short term drug exposure. The study performs intensive lab monitoring with a cross-over design to compare short courses of monotherapy and dual-therapy. This is an open-labeled study of a dual NRTI/NtRTI combination, ABC + TDF, compared to ABC and TDF monotherapy administered for 7 days. A screening genotype will be done to confirm that there are no resistance-associated mutations at baseline. Each subject will then be randomized to a 7-day sequence of monotherapy (ABC or TDF), and four measurements for plasma HIV RNA will be done to calculate the slope of the phase one viral decay. Prior to initiation of nucleoside analogues, PBMCs will be collected to measure baseline expression of nucleoside transport enzymes via RT-PCR and Western blot analysis. On days 7 and 8, serial blood specimens will be collected for plasma and intracellular levels of TDF and ABC. The monotherapy sequence will be followed by a 35-day washout period.

After the washout (day 42), subjects will initiate the dual NRTI/NtRTI therapy sequence for an additional 7 days. During dual NRTI/NtRTI therapy, again, four measurements for HIV RNA will be done to calculate the slope of the phase one viral decay. On day 48 and 49, serial plasma and intracellular levels of ABC + TDF will be evaluated. On Day 49 a second HIV genotype will be performed in real time. On day 49, after the second 7-day sequence, all subjects will receive EFV in addition to the ABC + TDF combination for 14 days. Afterwards, a second sample of PBMCs will be collected to evaluate for a potential induction or suppression of nucleoside transport enzymes. Since the long-term efficacy of the TDF + ABC nucleoside backbone is not yet known, TDF will be discontinued (day 63) and 3TC will be substituted. Subjects will then continue on the HAART portion of the study for an additional 46 weeks of EFV + ABC + 3TC.

ELIGIBILITY:
Inclusion Criteria:

1. HIV-1 infection, as documented by any licensed ELISA test kit and confirmed by Western blot at any time prior to study entry. HIV-1 culture, HIV-1 antigen, plasma HIV-1 RNA, or a second antibody test by a method other than ELISA is acceptable as an alternative confirmatory test.
2. Antiretroviral naïve defined as no prior therapy.
3. CD4+ cell count > than 200 cells/ mm3 determined by site clinical laboratory within 90 days of screening.
4. HIV-1 RNA level > 5000 copies/mL obtained by site clinical laboratory within 90 days of screening.
5. Laboratory values obtained by screening laboratories within 30 days of entry:

   * Absolute neutrophil count (ANC) ≥ 750/mm3.
   * Hemoglobin ≥ 8.0 g/dL.
   * Platelet count ≥ 50,000/mm3.
   * Calculated creatinine clearance (CrCl) > 50 mL/min as estimated by the
   * AST (SGOT), ALT (SGPT), and alkaline phosphatase ≤ 5 x ULN.
   * Total bilirubin ≤ 2.5 x ULN.
6. Negative serum or urine pregnancy test within 30 days of study entry.
7. Karnofsky performance score ≥ 70.
8. Men and women age ≥ 18 years.
9. Ability and willingness of subject to give written informed consent.

Exclusion Criteria:

1. Any NRTI or NNRTI-associated resistance mutations as defined by the updated International AIDS Society-USA (IAS-USA) mutation list.
2. Pregnancy and breast-feeding.
3. Active drug or alcohol use or dependence that, in the opinion of the investigator, would interfere with adherence to study requirements.
4. Urgent need to initiate antiretroviral therapy, as determined by the patient's primary provider.
5. Serious illness (requiring systemic treatment and/or hospitalization) until subject either completes therapy or is clinically stable on therapy, in the opinion of the investigator, for at least 14 days prior to study entry.
6. Use of any immunomodulator, HIV vaccine, or investigational therapy within 30 days of study entry.
7. Use of human growth hormone within 30 days prior to study entry.
8. Initiation of testosterone or anabolic steroids within 30 days prior to study entry. (Exception: Chronic replacement dosages in patient's with diagnosed hypogonadism is allowed)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2004-12-07 (Actual); Primary Completion 2008-06-26 (Actual); Study Completion 2010-04-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard H Haubrich, MD, Study Chair — University California San Diego; Miguel A Goicoechea, MD, Principal Investigator — University California San Diego
Locations (5):
- United States (5):
  - UCI, Irvine, California
  - USC, Los Angeles, California
  - University of California San Diego, San Diego, California
  - Santa Clara Valley Medical Center, San Jose, California
  - Harbor-UCLA Medical Center, Torrance, California

REFERENCES:
- [Result] Goicoechea M, Jain S, Bi L, Kemper C, Daar ES, Diamond C, Ha B, Flaherty J, Sun S, Richman D, Louie S, Haubrich R; California Collaborative Treatment Group. Abacavir and tenofovir disoproxil fumarate co-administration results in a nonadditive antiviral effect in HIV-1-infected patients. AIDS. 2010 Mar 13;24(5):707-16. doi: 10.1097/QAD.0b013e32833676eb. PMID 20087154
- See also: CCTG homepage — https://www.cctg.ucsd.edu

RESULTS

PARTICIPANT FLOW:
Groups:
- Tenofovir: Monotherapy tenofovir (300mg) for 7 days followed by a 35-day washout period then 7 days of ABC + TDF dual therapy
- Abacavir: Monotherapy abacavir (600mg) for 7 days followed by a 35-day washout period then 7 days of ABC + TDF dual therapy
Period: Overall Study
Arm/Group | Tenofovir | Abacavir
Started | 10 | 11
Completed | 10 | 11
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Tenofovir | Abacavir | Total
Number analyzed (Participants) | 10 | 11 | 21
Age, Continuous [Median (Full Range); unit: years] — Age range was not provided per arm, only the total age range provided.
  years | NA [NA to NA] — age range was collected for the total population and it is not possible separate data by Arm/Group | NA [NA to NA] — age range was collected for the total population and it is not possible separate data by Arm/Group | 37 [25 to 71]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 2 | 6
  Male | 6 | 9 | 15
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 6 | 8 | 14
  Black | 0 | 1 | 1
  Asian | 1 | 1 | 2
  American Indian | 2 | 0 | 2
  Other or unknown | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Change in Short-term Virologic Response
Description: Relative potencies of two monotherapy regimens (TDF alone vs. ABC alone) compared to the dual NRTI regimen of TDF+ABC as assessed by the short-term virologic response. (Change in HIV RNA copies/mL at baseline and day 7 for monotherapy, baseline and day 49 for dual therapy.)
Time Frame: 49 days
Population: Median monotherapy decay slopes compared to dual therapy decay slopes after addition of second antiviral agent.
Measure: Median (Full Range); unit: log(10) copies/mL per day
Groups:
- Tenofovir: Monotherapy tenofovir (300mg) for 7 days followed by a 35-day washout period then 7 days of TDF + ABC dual therapy
Arm/Group | Tenofovir | Abacavir
Number analyzed (Participants) | 10 | 11
log(10) copies/mL per day
  monotherapy | -.11 [-.16 to -.03] | -.15 [-.25 to -.04]
  dual therapy (combined TDF+ABC) | -.16 [-.20 to -0.07] | -.16 [-.26 to -.05]

2. Primary Outcome: Compare the Plasma Data of the Two Monotherapy Regimens to the Dual NRTI Regimen
Description: At day 49 of Sequence 2 a 24-hour post dose plasma sample should be collected and processed. All 7 samples from the sparse PK (time 0, 30-min, 1-hr, 2-hr, 3-hr, 6-hr and 24-hr post dose) should be sent overnight to appropriate off-site lab for analysis. Since the patient is on dual therapy and the each drug is measured in separate labs each PBMC samples should be split at each time-point with half of the samples shipped to Gilead and half shipped to USC (two separate shipments). ALL plasma samples should be sent to USC. Since samples have to be split we will need to collect double the blood for the intracellular (PBMC) PK:
  Blood volume (PBMC-plasma): 40 mL - each draw Blood volume (plasma only): 3 mL - each draw Blood volume: 169 mL- over 2 days
  Plasma NRTI and intracellular ddNTP concentrations were measured 7 days after treatment with ABC or TDF alone and were compared to levels obtained after 7 days of treatment with both drugs
Time Frame: 49 days
Population: Plasma NRTI concentrations were measured after 7 days on monotherapy and after 7 days on dual therapy
Measure: Median (Full Range); unit: (mcg/mL)*hr
Arm/Group | Tenofovir | Abacavir
Number analyzed (Participants) | 10 | 11
(mcg/mL)*hr
  monotherapy | 3.82 [1.74 to 7.96] | 12.54 [6.35 to 24.67]
  dual therapy | 4.09 [1.85 to 13.92] | 13.62 [7.44 to 58.29]

3. Secondary Outcome: Evaluate Change in Cellular Regulatory Enzymes Involved With Nucleoside Analogue Transport Across Cell Membranes as Assessed by RT-PCR of Specific mRNA Transcripts
Description: At day 1 and day 63 a PBMC sample for RT-PCR of nucleoside analogue transport enzymes (enzymes for efflux, influx) will be collected. The day 1 specimen should be stored and sent with day 8 PK specimens to USC. Day 63 specimen should be sent to USC after collection and processing.
  Blood volume: 20 mL Blood volume: 20 mL
Time Frame: Day 1 and Day 63
Measure: Median (Full Range); unit: fmol/10^6 cells
Arm/Group | Tenofovir | Abacavir
Number analyzed (Participants) | 10 | 11
fmol/10^6 cells
  dGTP concentrations | 4026 [NA to NA] — The median value was taken from Goicoechea et al (2010) and the dispersion data was not reported and original data can not be ascertained | 2464 [NA to NA] — The median value was taken from Goicoechea et al (2010) and the dispersion data was not reported and original data can not be ascertained
  dATP concentrations | 3238 [NA to NA] — The median value was taken from Goicoechea et al (2010) and the dispersion data was not reported and original data can not be ascertained | 3314 [NA to NA] — The median value was taken from Goicoechea et al (2010) and the dispersion data was not reported and original data can not be ascertained

4. Secondary Outcome: Determine Total Number of NRTI-associated Mutations After 7 Days of ABC or TDF Monotherapy or After 7 Days of Dual NRTI Therapy With ABC + TDF
Description: Subjects will be randomized to either TDF or ABC PO route for 7 days, which involves a fixed number of subjects. A sample size of 20 subjects (10 ABC and 10 TDF monotherapy and 20 ABC+TDF dual-therapy in HIV-positive patients). We determined the count of NRTI-associated mutations that emerged after 7 days of ABC or TDF monotherapy or after 7 days of dual NRTI therapy with ABC + TDF.
Time Frame: 7 days
Measure: Number; unit: mutations
Arm/Group | Tenofovir | Abacavir
Number analyzed (Participants) | 10 | 11
mutations | 0 | 0

5. Secondary Outcome: Compare the Relative Viral Potency of TDF Monotherapy Versus ABC Monotherapy
Description: Eligible patients will be randomized into two monotherapy arms (TDF and ABC) for a short (one week) viral dynamics and pharmacokinetics evaluation to determine their potency. After a one-month washout period, all patients will start a dual-therapy of ABC+TDF. Viral dynamics and pharmacokinetics of the dual-therapy will be evaluated during the first week of the treatment. EFV will be added to the regimen after one week of the dual-therapy administered. Relative potencies of two monotherapy regimens (TDF alone vs. ABC alone) assessed by the short-term virologic response. (Change in HIV RNA copies/mL at baseline and day 7 for monotherapy)
Time Frame: Baseline and day 7
Measure: Median (Full Range); unit: log(10) copies/mL per day
Arm/Group | Tenofovir | Abacavir
Number analyzed (Participants) | 10 | 11
log(10) copies/mL per day | -0.11 [-0.16 to -0.03] | -0.15 [-0.25 to -0.04]

6. Primary Outcome: Compare the Intracellular Pharmacokinetic (PK) Data of the Two Monotherapy Regimens to the Dual NRTI Regimen
Description: At day 49 of Sequence 2 a 24-hour post dose intracellular (PBMC) should be collected and processed. All 7 samples from the sparse PK (time 0, 30-min, 1-hr, 2-hr, 3-hr, 6-hr and 24-hr post dose) should be sent overnight to appropriate off-site lab for analysis. Since the patient is on dual therapy and the each drug is measured in separate labs each PBMC samples should be split at each time-point with half of the samples shipped to Gilead and half shipped to USC (two separate shipments). ALL intracellular (PBMC) samples should be sent to USC. Since samples have to be split we will need to collect double the blood for the intracellular (PBMC) PK:
  Blood volume (PBMC-plasma): 40 mL - each draw Blood volume (plasma only): 3 mL - each draw Blood volume: 169 mL- over 2 days
  Intracellular ddNTP concentrations were measured after 7 days on monotherapy and after 7 days on dual therapy
Time Frame: 49 days
Population: Intracellular ddNTP concentrations were measured after 7 days on monotherapy and after 7 days on dual therapy
Measure: Median (Full Range); unit: fmol/10^6 cells
Arm/Group | Tenofovir | Abacavir
Number analyzed (Participants) | 10 | 11
fmol/10^6 cells
  monotherapy | 49.3 [25.2 to 916.8] | 72.2 [19.3 to 503.8]
  dual therapy | 108.1 [42.4 to 508.4] | 80.9 [26.8 to 376]

ADVERSE EVENTS:
Time Frame: 14 months
Arm/Group | Tenofovir | Abacavir
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/11
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/11
Other Adverse Events (participants affected / at risk) | 0/10 | 0/11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2004-09-01): https://cdn.clinicaltrials.gov/large-docs/90/NCT00214890/Prot_SAP_000.pdf